CLINICAL TRIAL: NCT03639870
Title: A Prospective, Multicenter Clinical Investigation of the Glaukos® Trabecular Micro-Bypass System, Model iS3, in Subjects With Refractory Glaucoma
Brief Title: Investigation of the Glaukos® Trabecular Micro-Bypass System, Model iS3, in Subjects With Refractory Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INFI-106-G2W3 (GC-011)
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Glaucoma
Keywords: refractory
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: The iStent infinite Trabecular Micro-Bypass System Model iS3 is a sterile, single-use injector system that is pre-loaded with three G2-W stents, and is designed to deliver the stents into Schlemm's canal. The three G2-W stents are heparin-coated and manufactured from implant grade titanium.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Implant Group (Experimental): Qualified eyes with refractory glaucoma will be implanted unilaterally with the Glaukos® Trabecular Micro-Bypass System Model iS3 (three G2-W stents per study eye), and will be followed through 12 months postoperative.
  Interventions: Device: Model iS3 three-stent trabecular micro-bypass system

INTERVENTIONS:
Device: Model iS3 three-stent trabecular micro-bypass system — Provided in Arm/Group descriptions.
  Other Names: Implant Group

SUMMARY:
Prospective, multi-center, single-arm clinical trial to evaluate the safety and effectiveness of the Glaukos® Trabecular Micro-Bypass System Model iS3 (three stents per study eye) in subjects with refractory glaucoma.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single arm, open-label clinical trial of the iS3 system. Up to 65 qualified subjects will be implanted with three G2-W stents in one eye and will be followed for 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of refractory open-angle glaucoma (including pigmentary and pseudoexfoliative glaucoma) that is uncontrolled despite medical therapy and/or prior conventional incisional intraocular glaucoma surgeries.
* Phakic or pseudophakic.
* Males or females, 45 years of age or older.

Exclusion Criteria:

* Traumatic, uveitic, neovascular, or angle-closure; or glaucoma associated with vascular disorders.
* Active corneal inflammation or edema.
* Retinal disorders not associated with glaucoma.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2018-07-10 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Primary effectiveness endpoint | Month 12 postoperative
  The change in mean diurnal IOP from baseline at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Stephens, O.D., Study Chair — Glaukos Corporation
Locations (1):
- Glaucoma Associates of Tx, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No